

# Effect of core strength training on C-level difficulty movements of Wushu routine athletes

NCT number: 2021-323

Time: 8/21/2021

## Effect of core strength training on C-level difficulty movements of Wushu routine athletes

Dear Professor

Hello!

I am a doctoral student in Physical Education in UPM. This is an experimental research process on the impact of core strength training on the C- level difficulty of Competitive Wushu routines. The subjects were 18-22year old Wushu athletes. The data obtained from this survey are only for academic research. Therefore, investigators sincerely invite experts to score each stage of investigators experiment, help investigators do this experiment better. Thank you very much.

This paper designs the core strength training scheme based on the query and reference of relevant literature and the characteristics of C-level difficult movements of Wushu. The training plan of the experimental group includes three stages (weeks 1-3; weeks 4-9; and week 10-12). Each stage consists of different difficulty levels. The training program is divided into 6difficulty levels, and the specific training contents are as follows:

Part I: Difficulty Level of Core Strength Training. (Table 1)

Table 1 Content of 6 difficulty levels

| | | • |
|--------|------------|--------------------------|
| 6 | difficulty | Content |
| levels | | |
| Static | action | Mainly to strengthen the |
| under | steady | muscle endurance and |
| state | | waist and abdomen |
| | | strength of the body. |
| No | load | Mainly to strengthen the |
| moven | nent in | fast muscle strength and |
| steady | state | waist and abdomen |

| | strength of the body. |
|--------------------|----------------------------|
| Static action | Mainly to strengthen the |
| under unstable | muscle endurance of the |
| state | body and the strength of |
| | the deep muscles of the |
| | waist and abdomen. |
| <b>Movement</b> to | Mainly to strengthen the |
| overcome its | muscle explosive force |
| own resistance | and waist of the body in a |
| in an unstable | dynamic state Abdominal |
| state | control force. |
| Free strength | _ |
| exercise in | strength and coordination |
| unstable state | ability of the body in a |
| | dynamic state. |
| Core explosive | Mainly to strengthen the |
| power exercise | muscle speed and the |
| under unstable | explosive strength of the |
| conditions | waist and abdomen in the |
| | dynamic process of the |
| | body. |

Expert score: your evaluation of the six difficulty levels of students' experiment is (the full score is 10 points: 10 points for very applicable, 9 points for more applicable, 8 points for basic applicable and 7 points for not applicable.):

| _ | 1 1 · |
|-----------------|-------------------------------|
| $\bigcirc$ Ve | ry applicable (10 points) |
| $\bigcirc_{Mc}$ | re applicable (9 points) |
| $\bigcirc$ Bas | sically applicable (8 points) |
| $\bigcirc_{No}$ | t applicable (7 points) |
| Modif | ication oninions of experts: |

### Part II: Core Strength Training Plan. (Weeks 1-3; weeks 4-9; and weeks 10-12)

(1) Basic stage of core strength training

Training time: 30 minutes three times a week for 1-3 weeks

Training content: static action in stable state, no-load movement in

stable state and static action in unstable state

Number and times of training groups (Table 2)

Table 2 contents of core strength training in week 1-3 basic stage

| Training Phase | Training Content | Time And |
|---|---|---|
| | | Frequency |
| Preparation part (5 minutes) | Jogging | 3 minutes 3×50m |
| | Neck movement (front, | 30S 4×8 |
| | rear, left and right) | |
| | Shoulder movement | 30S 4×8 |
| | Waist movement | 30S 4×8 |
| | Lunge leg press | 30S 4×8 |
| Static action under steady | Flat brace | 60S × 2 groups |
| state (12 minutes) | | |
| | Single side support of | $60S \times 2$ groups |
| | flat support (left) | |
| | Single side support of | $60S \times 2$ groups |
| | flat support (right) | |
| | Reverse plate support | $60S \times 2$ groups |
| | Side bridge elbow | 60S × 2 groups |
| | support (left) | |
| | Side bridge elbow | 60S × 2 groups |
| | support (right) | |
| No load movement in | Suspension leg lift | 60S × 3 groups |
| steady state (9 minutes) | | |
| | Drape knees and tuck | 60S × 2 groups |
| | in (left) | |

| | Drape, 1 | bend | knees and | 60S × 2 groups |
|---|---|---|---|---|
| | tuck in ( | right | <u>:</u> ) | |
| | Hanging | g ups | ide down | 60S × 2 groups |
| Static action under unstable | Lateral | hip | abduction | $60S \times 2$ groups |
| state (4 minutes) | (left) | | | |
| | Lateral | hip | abduction | 60S × 2 groups |
| | (right) | | | |

| Expert score: your evaluation of the content and structure of the |
|-----------------------------------------------------------------------------|
| students' experiment in the first stage is (the full score is 10 points, 10 |
| points are very applicable, 9 points are more applicable, 8 points are |
| basically applicable, and 7 points are not applicable.) |
| OVery applicable (10 points) |
| O More applicable (9 points) |
| OBasically applicable (8 points) |
| ONot applicable (7 points) |
| Modification opinions of experts: |

### (2) Core strength training consolidation stage

Training time: 30 minutes three times a week for 4-9 weeks

Training content: Static action in unstable state, movement to overcome self-resistance in unstable state, free force exercise in unstable state.

Number and times of training groups (Table 3)

Table 3 contents of core strength training in week 4-9 basic stage

| Training Phase | Training Content | Time And |
|------------------------------|-----------------------|-----------------|
| | | Frequency |
| Preparation part (6 minutes) | Jogging | 4 minutes 4×50m |
| | Neck movement (front, | 30S 4×8 |
| | rear, left and right) | |
| | Shoulder movement | 30S 4×8 |
| | Waist movement | 30S 4×8 |

| | Lunge leg press | 30S 4×8 |
|---|---|---|
| Static action under unstable | Lateral hip abduction | 60S ×3groups |
| state (6 minutes) | (left) | |
| | Lateral hip abduction | $60S \times 3$ groups |
| | (right) | |
| Movement to overcome its | Push down leg arm flat | 60S × 3 groups |
| own resistance in an | hip (left) | |
| unstable state (9 minutes) | | |
| | Push down leg arm flat | 60S ×3groups |
| | hip (right) | |
| | Upside down | 60S ×3 groups |
| | abdominal retraction | |
| | (bilateral) | |
| Free strength exercise in | Prone mass body | 60S × 3groups |
| unstable state (9 minutes) | | |
| | Prone push-pull | 60S × 3 groups |
| | Swiss Ball push up | 60S × 3 groups |

Expert score: your evaluation of the content and structure of the students' experiment in the second stage is (the full score is 10 points, 10 points are very applicable, 9 points are more applicable, 8 points are basically applicable, and 7 points are not applicable.)

| O Very applicable (10 points) |
|-----------------------------------|
| O More applicable (9 points) |
| OBasically applicable (8 points) |
| O Not applicable (7 points) |
| Modification opinions of experts: |

#### (3) Core strength training improvement stage

Training time: 30 minutes three times a week for 10-12 weeks
Training contents: free strength exercise under unstable conditions,
core explosive force exercise under unstable conditions, and core

special strength exercise under unstable conditions.

Number and times of training groups (Table 4)

Table 4 contents of core strength training in week 4-9 basic stage

| Training Phase | Training Content | Time And |
|------------------------------|-------------------------|-----------------|
| | | Frequency |
| Preparation part (4 minutes) | Jogging | 2 minutes 2×50m |
| | Neck movement (front, | 30S 4×8 |
| | rear, left and right) | |
| | Shoulder movement | 30S 4×8 |
| | Waist movement | 30S 4×8 |
| | Lunge leg press | 30S 4×8 |
| Free strength exercise in | Flat brace (two points) | 60S × 2groups |
| unstable state (10 minutes) | Prone mass body | 60S ×2groups |
| | Prone push-pull | 60S ×2 groups |
| | Swiss Ball push up | 60S × 4 groups |
| No load movement in | Suspension leg lift | 60S × 2 groups |
| steady state (8 minutes) | Drape knees and tuck | 60S × 2 groups |
| | in (left) | |
| | Drape, bend knees and | 60S × 2 groups |
| | tuck in (right) | |
| | Hanging upside down | 60S × 2groups |
| Core explosive force | Lie on your back and | 60S × 2 groups |
| exercise under non-stability | bend your knees at | |
| (8minutes) | both ends | |

| Plate support knee lift | 60S × 2 groups |
|--------------------------|----------------|
| Rotation of stretch belt | 60S × 2 groups |
| (both sides) | |
| Lie on your back and | 60S × 2 groups |
| throw the ball | |

| Expert score: your evaluation of the content and structure of the |
|---------------------------------------------------------------------------|
| students' experiment in the second stage is (the full score is 10 points, |
| 10 points are very applicable, 9 points are more applicable, 8 points are |
| basically applicable, and 7 points are not applicable.) |
| Warranniachla (10 nainta) |

| OVery applicable (10 pe | points) |
|-------------------------|---------|
|-------------------------|---------|

- O More applicable (9 points)
  O Basically applicable (8 points)
  O Not applicable (7 points)

Modification opinions of experts: